CLINICAL TRIAL: NCT02662556
Title: A Multicenter, Open-Label Trial to Evaluate the Safety and Efficacy of the Sufentanil Sublingual Tablet 30 mcg in Patients With Post-Operative Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Talphera, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAP303
Record Dates: First submitted 2016-01-20; First posted 2016-01-25 (Estimated); Results first posted 2017-03-15 (Actual); Last update posted 2017-03-15 (Actual); Status verified 2017-01

CONDITIONS: Acute Moderate-to-severe Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- sufentanil sublingual tablet 30 mcg (Experimental): sufentanil sublingual tablet 30 mcg
  Interventions: Drug: sufentanil sublingual tablet 30 mcg

INTERVENTIONS:
Drug: sufentanil sublingual tablet 30 mcg — sufentanil sublingual tablet 30 mcg as needed for pain management, but no more frequently than every 60 minutes, for up to 12 hours.
  Other Names: ST 30 mcg

SUMMARY:
This is a multicenter, open-label study in patients 40 years and older who are undergoing a surgical procedure.

Patients may receive one dose of ST 30 mcg as needed for pain management, but no more frequently than every 60 minutes, for up to 12 hours.

DETAILED DESCRIPTION:
This is a multicenter, open-label study in patients 40 years and older who are undergoing a surgical procedure.

Upon meeting all entrance criteria, patients will be administered the first dose of ST 30 mcg and will remain in the study for up to 12 hours for safety and efficacy measurements. Patients may receive additional doses of ST 30 mcg as needed for pain management, but no more frequently than every 60 minutes.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients who are 40 years of age or older.
2. Patients who have undergone a surgical procedure with general anesthesia or spinal anesthesia that does not include intrathecal opioids during the operation.
3. Patients classified as American Society of Anesthesiologists (ASA) class IIII (Appendix I).

Exclusion Criteria:

1. Patients who have taken an opioid for more than 30 consecutive days, at a daily dose of more than 15 mg of morphine (or equivalent), within the past 3 months prior to surgery (e.g. more than 3 doses per day of Vicodin®, Norco®, Lortab® with 5 mg hydrocodone per tablet).
2. Patients with a positive drug of abuse screen unless the positive test result is consistent with a prescribed medication.
3. Patients with a history of opioid dependence within 2 years before the start of the study, defined as meeting the DSM-IV-TR™ Criteria for Substance Dependence specified in Appendix II.
4. Patients who have used any illicit drugs of abuse within five years before the start of the study.
5. Patients who have abused any prescription medication or alcohol within one year before the start of the study.
6. Patients with an allergy or hypersensitivity to opioids.
7. Patients who are currently taking monoamine oxidase inhibitors (MAOIs) or have taken MAOIs within 14 days of the first dose of study drug.
8. Patients with current sleep apnea that has been documented by a sleep laboratory study or are on home continuous positive airway pressure (CPAP).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2016-03; Primary Completion 2016-06 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela P. Palmer, MD, PhD, Study Director — Talphera, Inc
Locations (2):
- United States (2):
  - HD Research, Houston, Texas
  - Research Concepts, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Sufentanil Sublingual Tablet (SST) 30 mcg: Sufentanil sublingual tablet (SST) 30 mcg
  Sufentanil sublingual tablet (SST) 30 mcg: sufentanil sublingual tablet 30 mcg as needed for pain management, but no more frequently than every 60 minutes, for up to 12 hours.
Period: Overall Study
Arm/Group | Sufentanil Sublingual Tablet (SST) 30 mcg
Started | 140
Completed | 132
Not Completed | 8
Not completed — Adverse Event | 4
Not completed — Lack of Efficacy | 4

BASELINE CHARACTERISTICS:
Arm/Group | Sufentanil Sublingual Tablet (SST) 30 mcg
Number analyzed (Participants) | 140
Age, Categorical [Count of Participants; unit: Participants] — All subjects must have been at least 40 years of age at the time of screening
  Participants
    <=18 years | 0
    Between 18 and 65 years | 116
    >=65 years | 24
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75
  Male | 65

OUTCOME MEASURES:

1. Primary Outcome: Time-weighted Summed Pain Intensity Difference (SPID) Over the 12-hour Study Period (SPID12).
Description: The pain intensity difference (PID) at each evaluation time point after the dose of study drug is the difference in pain intensity at the specific evaluation time point and baseline pain intensity [PID(evaluation time after the first dose) = PI(baseline) - PI(evaluation time after the first dose)]. A pain intensity score ranging from 0 (no pain) to 10 (worst possible pain) is obtained at baseline and throughout the 12 hour period. The time-weighted SPID12 is the time-weighted summed PID over the 12-hour study period. The scores ranged from -13.75 to 100.5. A negative score indicates an increase in pain intensity and a higher score indicates a greater decrease in pain intensity.
Time Frame: 12-hours
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Sufentanil Sublingual Tablet (SST) 30 mcg: Sufentanil sublingual tablet (SST) 30 mcg
  Sufentanil sublingual tablet (SST) 30 mcg: one sufentanil sublingual tablet 30 mcg as needed for pain management, but no more frequently than every 60 minutes, for up to 12 hours.
Arm/Group | Sufentanil Sublingual Tablet (SST) 30 mcg
Number analyzed (Participants) | 137
units on a scale | 36.04 (2.22)

2. Secondary Outcome: Time-weighted Summed Pain Intensity Difference (SPID) Over the First Hour (SPID1).
Description: The pain intensity difference (PID) at each evaluation time point after the dose of study drug is the difference in pain intensity at the specific evaluation time point and baseline pain intensity [PID(evaluation time after the first dose) = PI(baseline) - PI(evaluation time after the first dose)]. A pain intensity score ranging from 0 (no pain) to 10 (worst possible pain) is obtained at baseline and throughout the 1 hour period. The time-weighted SPID1 is the time-weighted summed PID over the 1-hour study period. The scores ranged from -6.67 to 6.77. A negative score indicates an increase in pain intensity and a higher score indicates a greater decrease in pain intensity.
Time Frame: 1 hours
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Sufentanil Sublingual Tablet (SST) 30 mcg
Number analyzed (Participants) | 137
units on a scale | 0.87 (0.16)

3. Secondary Outcome: Percentage of Patients Who Responded to the Global Assessments as "Excellent" or "Good"
Description: Patients were asked "Overall, how would you rate the method of pain control"? Poor (1), Fair (2), Good (3), or Excellent (4)
Time Frame: 12 hours or at patients' termination from study
Population: 135 patients completed the scale
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Sufentanil Sublingual Tablet (SST) 30 mcg
Number analyzed (Participants) | 135
percentage of subjects | 87.4 [81.81 to 93.00]

4. Secondary Outcome: Percentage of Healthcare Professionals Who Responded to the Global Assessments as "Excellent" or "Good"
Description: Healthcare professionals were asked "Overall, how would you rate the method of pain control"? Poor (1) Fair (2) Good (3) Excellent (4)
Time Frame: 12 hours or until patients' termination from study
Measure: Number (95% Confidence Interval); unit: percentage of healthcare professionals
Arm/Group | Sufentanil Sublingual Tablet (SST) 30 mcg
Number analyzed (Participants) | 123
percentage of healthcare professionals | 90.2 [85.00 to 95.49]

ADVERSE EVENTS:
Time Frame: Spontaneous reports throughout patients' participation in study through study completion.
Description: SAEs were reported if occurrence was within 30 days of last dose of study medication.
Arm/Group | Sufentanil Sublingual Tablet (SST) 30 mcg
Serious Adverse Events (participants affected / at risk) | 1/140
Other Adverse Events (participants affected / at risk) | 45/140
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sufentanil Sublingual Tablet (SST) 30 mcg (N=140)
Acute Stroke (Nervous system disorders) | 1 (1) — Occurred after patient's participation in study; Deemed unrelated to study drug
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sufentanil Sublingual Tablet (SST) 30 mcg (N=140)
Nausea (Gastrointestinal disorders) | 38 — Events entered in the list were noted as possibly or probably related to study drug
Dizziness (Nervous system disorders) | 6
Headache (Nervous system disorders) | 4
Pruritis (Skin and subcutaneous tissue disorders) | 4
Oxygen saturation decreased (Investigations) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other